CLINICAL TRIAL: NCT03250195
Title: Non-invasive Detection of Male Infertility With FDG-PET/MRI (Spectroscopy and DWI)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient inclusion of patients
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Louise Madeleine Risør, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-17013319
Record Dates: First submitted 2017-08-07; First posted 2017-08-15 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Fertility Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/MRI (Other): All participants will have a PET/MRI performed
  Interventions: Diagnostic Test: PET/MRI

INTERVENTIONS:
Diagnostic Test: PET/MRI — PET/MRI scan

SUMMARY:
The aim of the study is to examine the value of the new MRI techniques (spectroscopy and DWI), and FDG-PET in prognostication of male infertility.

DETAILED DESCRIPTION:
The diagnostic workup of male infertility includes medical history, physical examination and semen analysis. In severe cases further workup includes testicular ultrasound, analysis of genes and hormones and in a few cases testicular biopsies are necessary.

Ultrasound is the first choice of imaging, but new MRI and PET techniques can provide additional information.

Research indicates that new MRI techniques can measure the activity of the testicular sperm cell production non-invasively and FDG-PET can measure the testicular metabolism with a radioactively marked glucose analog (FDG). These imaging modalities are combined in a PET/MRI and we wish to perform a PET/MRI in 10 men with normal sperm counts and 10 men with low sperm counts in order to evaluate whether a PET/MRI can distinguish testicles with and without sperm cell production. We hope that this new non-invasive technique can replace the need for invasive biopsies and will be able to target the harvesting of sperm cells in fertility treatment.

ELIGIBILITY:
Inclusion Criteria:

18-40 year old males referred to fertility treatment at Rigshospitalet, Denmark. 10 men with a normal sperm count and 10 men with no sperm cells in the ejaculate will be included. The patients shall be able to understand the patient information and be able to give informed consent.

Exclusion Criteria:

Severe claustrophobia Age: less than 18 or above 40 Severe obesity (> 140 kg) Pacemaker or other electronic in-operated devices Non-MR compatible metallic devices Malignant testicular tumors suspected at clinical examination or ultrasound Infectious testicular diseases

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We examine testicular function and therefore we only include men
Enrollment: 12 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2021-08-07 (Actual); Study Completion 2021-08-07 (Actual)

PRIMARY OUTCOMES:
SUVmax (maximum standardized uptake value) | 1 year
  The SUV is the ratio of the image derived radioactivity concentration and the whole body concentration of the injected radioactivity.
Testicular metabolite concentrations measured by MRI spectroscopy. | 1 year
  MR spectroscopy is a non-invasive, ionizing-radiation-free analytical technique that has been used to study metabolic changes in different tissues. The unit is p.p.m.
Testicular apparent diffusion coefficient | 1 year
  Diffusion-weighted magnetic resonance imaging (DW MRI) provides image contrast that is dependent on the random microscopic motion of water protons, which may be substantially altered by different pathological process.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Risør, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Østerbro, Denmark

IPD SHARING:
Plan to Share IPD: No
The results will be published in international journals